CLINICAL TRIAL: NCT07320404
Title: Arthroscopic Scaphoid Bone Graft Combined With Percutaneous Fixation Versus Open Scaphoid Fixation With Non Vascularized Graft in Scaphoid Non-union
Brief Title: Arthroscopic Scaphoid Grafting Versus Open Grafting in Scaphoid Non Union
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAMSU MD 288/2019
Record Dates: First submitted 2024-07-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-07

CONDITIONS: Scaphoid Fracture Non Union

STUDY DESIGN:
Intervention Model Description: 2 groups one with the arthroscopic grafting combined with percutaneous fixation, the second with opend grafting and fixation by K wires.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arthroscopic A group (Experimental): arthroscopic bone grafting combined with percutaneous K wires fixation for scaphoid non union patients
  Interventions: Procedure: Arthroscopic grafting and k wires fixation
- open O group (Experimental): open volar or dorsal scaphoid grafting with K wires fixation for scaphoid non union patients
  Interventions: Procedure: open scaphoid grafting with K wires fixation

INTERVENTIONS:
Procedure: Arthroscopic grafting and k wires fixation — Arthroscopic midrcarpal scaphoid non union debridment and iliac cancellous bone grafting with K wires fixation
  Arms: arthroscopic A group
Procedure: open scaphoid grafting with K wires fixation — open surgical volar or dorsal scaphoid non union site debridment and application of iliac bone graft and K wires fixation
  Arms: open O group

SUMMARY:
the investigators compare the arthroscopic grafting technique with the traditional open technique in th treatment of scaphoid non union as regards the union rate, time to union and functional outcomes to provide the best intervention to the patient

DETAILED DESCRIPTION:
The treatment of scaphoid non union has no gold standard technique so in this study the investigators try to compare the arthroscopic and the open grafting techniques to determine the better technique to achieve union, time to union and the better functional outcomes including wrist range of motion and grip strength as a primary outcome and the secondary outcomes are the operative time, the complications and radiological correction of the hum-back deformity if present.

ELIGIBILITY:
Inclusion Criteria:

* scaphoid non-union cases
* 16 years or older
* males or females
* independent from chronicity or non-union location and the investigators defined the non union as failure to reach scaphoid union up to 6 months

Exclusion Criteria:

.Revision scaphoid non-union cases.

* Previously operated wrist for any other pathology
* Avascular necrosis (AVN) confirmed by intraoperative inspection.
* Scaphoid non-union advanced collapse (SNAC) stage 2 and higher.
* Any associated wrist pathology that required separate treatment surgical approach.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
union rate | 6 months
  percentage of patients in each arm that achieve bony union
time to union | 6 to 24 weeks
  the time that patient take to achieve bony union
wrist flexion and extension | preoperative, at 6 months and at 24 months
  flexion and extension range of motion
wrist radial and ulnar deviation | preoperative, at 6 months and at 24 months
  radial and ulnar deviation range of motion
grip strength | preoperative , at 6 months and at 24 months
  the power of hand grip measured by dynamometer
The disability of arm, shoulder and hand score (DASH score) | preoperative , at 6 months and at 24 months
  a questionnaire to assess upper limb function from 0 to 100 where the lower the score means better outcome
The Mayo modified wrist score | preoperative, at 6 months and at 24 months
  A functional score that depends on the patients function and examination from 0 to 100 and the higher the score the higher the outcome

SECONDARY OUTCOMES:
complications | 2 years post operative
Degree of scaphoid hump back deformity correction | post operative after bony union up to 1 year
  Radiological parameter thorough scapholunate angle
Operative time | intraoperative
  the duration of each operation

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed El-Mahy, prof., Study Chair — Ain Shams University
Locations (1):
- Faculty of medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jegal M, Kim JS, Kim JP. Arthroscopic Management of Scaphoid Nonunions. Hand Surg. 2015;20(2):215-21. doi: 10.1142/S0218810415400031. PMID 26051763
- [Result] Munk B, Larsen CF. Bone grafting the scaphoid nonunion: a systematic review of 147 publications including 5,246 cases of scaphoid nonunion. Acta Orthop Scand. 2004 Oct;75(5):618-29. doi: 10.1080/00016470410001529. PMID 15513497